CLINICAL TRIAL: NCT04385927
Title: Life Beyond Trauma: 1-on-1 e-Health Program for Parents of Neurodiverse Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Child-Bright Network (Other)
Responsible Party: Principal Investigator, Patrick J. McGrath, Principal Investigator, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23865
Record Dates: First submitted 2020-03-23; First posted 2020-05-13 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Post Traumatic Stress Injury; Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate e-NET Group (Experimental): Parents of neurodiverse children with PTSI will receive e-NET immediately after the baseline survey
  Interventions: Behavioral: e-Net for Parents of Neurodiverse Children
- Wait List Control Group (Experimental): Parents of neurodiverse children with PTSI will receive e-NET 3 months after the baseline survey
  Interventions: Behavioral: e-Net for Parents of Neurodiverse Children

INTERVENTIONS:
Behavioral: e-Net for Parents of Neurodiverse Children — One-on-one distance coached intervention; approx. 12 sessions at 60-90 minutes.

SUMMARY:
Parents of neurodiverse children are more likely to experience traumatic events related to the care of their child/children. This increases the probability to experience Posttraumatic Stress Injury (PTSI). However, interventions addressing PTSI symptoms in parents are rare.

In this research project the study investigators will test the feasibility and efficacy of e-NET, a distance-delivered, exposure-based intervention for PTSI adapted to the needs of parents of neurodiverse children. E-NET is an adapted version of the Narrative Exposure Therapy (NET), an evidence-based intervention approach for individuals with PTSI who have experienced repeated or continuous trauma. The intervention will be conducted via videoconferencing with trained paraprofessionals. During the intervention a narrative of both positive and negative (traumatic) experiences in the parents' life will be created. The intervention contains approx. 12 one-on-one sessions with a trained paraprofessional via videoconferencing.

The study design is a waitlist control group design. Approx. 20 participants will receive e-NET directly after the baseline survey and 20 participants will receive e-NET approx. 3 months after the baseline survey. To test the efficacy of the intervention, participants will fill out surveys about PTSI and other mental health symptoms before, directly after, and 2 and 6 months after the intervention. Adverse events and distress will be assessed in every session. As part of the baseline, participants will complete the survey "Surviving and Thriving in Parenting Neurodiverse Children" to determine their eligibility for the intervention. Main eligibility criterion is the presence of PTSI symptoms.

ELIGIBILITY:
Inclusion Criteria: Parent/Caregivers must meet the following criteria to be eligible to move on to Consent

1. Be a parent/caregiver of a neurodiverse child
2. Be at least 18 years of age
3. Be able to understand spoken and written English at a Grade 8 level
4. Fulfill the criteria of full or subclinical PTSI according to DSM-5, measured with the Life Events Checklist for DSM-5, the Parent Trauma Checklist and the PTSD Checklist for DSM-5. For this they have to report at least one traumatic event in the LEC-5 or the Stressful Life Experiences of Parents Checklist. To fulfill all PTSI criteria, the participant additionally needs to respond with "moderately" or higher in at least one item for the criteria B and C and two items for criteria D and E. Subclinical PTSI is fulfilled if the participant meets all but one criterion of B, C, D, or E is not met.
5. Have access to a computer with high speed Internet
6. Live in Canada
7. Commit to the requirements of taking part in the study (12 weekly coaching calls)

Exclusion Criteria:

1. Acute suicidal behavior or other extreme forms of self-destructive behavior
2. Moderate to severe symptoms of dissociation
3. Acute psychotic symptoms
4. Previously participated in exposure intervention for PTSI/PTSD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in PTSI symptoms | Baseline, Immediately Post- intervention, 2 months post-intervention, 6 months post-intervention
  PTSD symptoms are measured with the PTSD Checklist - 5 (PCL-5). Respondents are asked to rate how bothered they have been by each of 20 items in the past month on a 5- point Likert scale ranging from 0-4. Items are summed to provide a total severity score. Higher scores indicate a worse outcome

SECONDARY OUTCOMES:
Change in Overall Health | Baseline, Wait-list Baseline; through study completion, an average of 12 weeks; Immediately Post-assessment; 2 month follow up; 6 month follow up
  General health will be measured with the questionnaire PROMIS Global Health Caregiver's general health
Change in Depression Symptoms | Baseline, Immediately Post-assessment, 2 month follow up, 6 month follow up
  Depression symptoms will be measured with the Patient Health Questionnaire (PHQ-9)
Change in overall functionality | Baseline; Wait list Baseline, Immediately Post intervention; 2 month follow up; 6 month follow up
  Functionality will be measured with the Sheehan Disability Scale (SDS). SDS is measured on a 10-point scale (0-9). Higher score indicates a worse outcome.
Posttraumatic Growth | Baeline; Wait list Baseline; Immediately Post intervention; 2 month follow up; 6 month follow up
  Posttraumatic growth will be measures using the Posttraumatic Growth Inventory - Short Form (PTGI ). The PTGI is measured on a 6-point Likert scale (score 0-5). Higher score indicates a better outcome.
Parent-child Relationship | Baseline; Wait list Baseline; Immediately Post intervention; 2 month follow up; 6 month follow up
  The parent-child relationship will be measured with the Parent and Family Adjustment Scales (PAFAS). Items are rated from 0 to 3. Note that shaded items in the scoring key below must be reverse scored (i.e. 0=3, 1=2, 2=1, 3=0) before summing the Total Score. High scores indicate worse outcome.
Satisfaction with Lifeline Tool | During week 1 of intervention
  The satisfaction with Lifeline Tool (self-constructed) will be measured with a self-constructed 3-item usability questionnaire. It is scored on a five point scale. Items are rated from 0-4. Higher score indicates better outcome.
Change in Anxiety Symptoms | Baseline, Immediately Post-assessment, 2 month follow up, 6 month follow up
  Anxiety Symptoms are measured with the Generalized Anxiety Disorder (GAD-7). Items are scored on a four point scale, items are rated from 0-3. Higher score indicates better outcome.
Change in Physical Health Symptoms | Baseline; throughout study completion, approximately 12 week; Immediately Post-assessment; 2 month follow up; 6 month follow up
  Physical Health symptoms will be assessed with the Patient Health Questionnaire Physical Symptoms (PHQ-15). Items are scored on a three point scale, items are rated from 0-2. Higher score indicates worse outcome.
Adverse Events | throughout study completion, approximately 12 weeks; immediately post intervention
  Adverse events will be assessed with a self-constructed questionnaire for adverse events, the course of symptoms during intervention and general distress.
Therapeutic Alliance | Immediately post intervention
  The interaction between coach and client will be assessed through the Therapeutic Alliance- Working Alliance Inventory - Short Form Revised (WAI-SR)
Participant Satisfaction | Immediately Post intervention
  Client satisfaction will be assessed with the Client Satisfaction Questionnaire (CSQ-8) and some additional (self-constructed) qualitative questions. CAQ-8 Items are scored on a four point scale, items are rated from 0-3. Higher score indicates worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick McGrath, PhD, Principal Investigator — IWK Health Centre; Elisa Kaltenbach, PhD, Principal Investigator — IWK Health Centre
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jones KA, Freijah I, Brennan SE, McKenzie JE, Bright TM, Fiolet R, Kamitsis I, Reid C, Davis E, Andrews S, Muzik M, Segal L, Herrman H, Chamberlain C. Interventions from pregnancy to two years after birth for parents experiencing complex post-traumatic stress disorder and/or with childhood experience of maltreatment. Cochrane Database Syst Rev. 2023 May 4;5(5):CD014874. doi: 10.1002/14651858.CD014874.pub2. PMID 37146219
- [Derived] Kaltenbach E, Chisholm M, Xiong T, Thomson D, Crombach A, McGrath PJ. Online narrative exposure therapy for parents of children with neurodevelopmental disabilities suffering from posttraumatic stress symptoms - study protocol of a randomized controlled trial. Eur J Psychotraumatol. 2021 Nov 21;12(1):1991650. doi: 10.1080/20008198.2021.1991650. eCollection 2021. PMID 34868484